CLINICAL TRIAL: NCT07355621
Title: A Single-center, Randomized, Double-blind, Placebo-controlled Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of UP-818-CC Injection in Healthy Chinese Subjects After Single-dose and Multiple-dose Intravenous Infusion
Brief Title: UP-818-CC Injection in Healthy Chinese Subjects
Acronym: UP-818-CC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EnliTISA (Shanghai) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UP-19-818-21002
Record Dates: First submitted 2025-12-07; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Healthy Subjects
Keywords: UP-818-CC injection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP-818-CC group (Experimental): single or multiple intravenous UP-818-CC injection
  Interventions: Drug: UP-818-CC injection
- placebo group (Placebo Comparator): single or multiple intravenous placebo injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UP-818-CC injection — UP-818-CC injection
  Arms: UP-818-CC group
Other: Placebo — placebo
  Arms: placebo group

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability and pharmacokinetic characteristics in healthy Chinese volunteers after single and multiple dose of intravenous infusion of UP-818-CC.

This study is divided into two parts, single ascending dose part (SAD) and multiple ascending dose part (MAD), both conducted in healthy subjects, using a randomized, double-blind, placebo-controlled, dose-escalating design.

The SAD part is planned to be carried out in 6 dose groups. A total of about 43 healthy adult subjects are planned to be included. All subjects will receive a single dose on the first day (D1).

According to the obtained PK and safety information of the SAD, three appropriate dose groups are selected in MAD. A total of about 30 healthy adult subjects, both male and female, will be included. All subjects will receive multiple doses from D1 to D7, once daily.

ELIGIBILITY:
Inclusion Criteria:

1. Male weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) in the range of 19 to 26, including boundary values, BMI = weight (kg) / height (m) 2;
2. The medical history, physical examination, laboratory items and tests related to the trial are all normal or abnormal and have no clinical significance, and the clinical research doctor judges that they are qualified;
3. During the trial and within 3 months after the trial, the subjects or their spouses voluntarily took effective contraceptive measures, such as abstinence, condoms, the use of intrauterine devices, double-barrier methods (such as condoms and contraceptive diaphragms), etc., female subjects enter the trial after confirming the menstrual period; male subjects have no sperm donation plan;
4. Be able to communicate well with researchers, fully understand the purpose and requirements of this trial, voluntarily participate in clinical trials and sign written informed consent.

Exclusion Criteria:

1. Those who are allergic to any active ingredient of the investigational drug or any excipient or excipient;
2. Allergies (including bronchial asthma or asthmatic bronchitis, allergic rhinitis and other multiple drug or food allergies, etc.) or the total IgE results of the screening period showed allergies;
3. Those with past or current diseases that the investigator considers ineligible to enroll, including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, genitourinary system, metabolism and bone, or those with a history of allergic diseases or malignant tumors;
4. Past or current chronic obstructive pulmonary disease, active pulmonary tuberculosis (including but not limited to increased erythrocyte sedimentation rate or a positive T-cell spot test for tuberculosis infection in the screening period or abnormal and clinically significant chest CT examination in the screening period, judged by the investigator afterwards, only those with calcifications and no clinically significant symptoms on lung imaging examinations can be enrolled) and other respiratory diseases;
5. Patients with acute infection within 2 weeks before screening;
6. Difficulty in venous blood collection, or those with a history of needle dizziness or haemorrhage;
7. Frequent excessive consumption of tea, coffee or caffeinated beverages (more than 8 cups a day, 1 cup = 200 ml) in the 3 months prior to screening or ingestion of any food or drink containing caffeine, alcohol, xanthine or grapefruit within 48 hours prior to randomization;
8. History of binge drinking or frequent alcohol consumption within 6 months prior to the trial (more than 14 units of alcohol per week, 1 unit = 360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine) or alcohol breath test the day before dosing is positive (breath alcohol content > 0.0 mg/100 mL), or those who cannot abstain from alcohol during the test;
9. Those who have participated in any drug clinical trial and have taken the investigational drug within 3 months before screening;
10. Donate blood or lose ≥400 mL of blood within 3 months before screening (except for female menstrual blood loss), or plan to donate blood or blood components during the study or within 3 months after the end of the study;
11. Persons with a history of drug abuse/dependence or drug history within 1 year before screening, or those with positive drug abuse screening (screening items may include: morphine, THC, methamphetamine, DMD fetamine, ketamine and cocaine);
12. Those who smoked more than 5 cigarettes per day within 3 months before screening and those who could not smoke during the whole trial period;
13. Have used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, etc.) or health products within 14 days before screening;
14. Post-vaccination within 4 weeks prior to the first dose of investigational drug or planned within 4 weeks after the last dose is discontinued, live vaccines including but not limited to: measles, mumps, rubella, chickenpox, yellow fever, rabies, BCG Bacillus, typhoid vaccine, live COVID-19 vaccine, etc.;
15. During the screening period, the QTcF interval >450 milliseconds (msec) or the abnormal and clinically significant results of the 12-lead ECG;
16. During the screening period, the investigators determined that the vital signs were abnormal: systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <50 mmHg or ≥90 mmHg, or the body temperature, heart rate, pulse, respiration, blood oxygen saturation and other indicators exceeded the center normal value range and the investigator judges that the abnormality has clinical significance;
17. During the screening period, estimated glomerular filtration rate (eGFR) <90 mL/min/1.73 m2 by MDRD equation (Appendix 3);
18. Those who are positive for one or more of hepatitis B surface antigen, hepatitis C virus (HCV) antibody, syphilis antibody (TPPA) or human immunodeficiency virus (HIV) antibody;
19. Those who cannot communicate or cooperate with medical staff due to neurological, mental illness or language barriers;
20. The investigator believes that the subjects are not suitable to participate in the trial, or the subjects cannot participate in the trial due to their own reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as coded by MedDRA and assessed by CTCAE v5.0 | From baseline to Day4 in single dose groups, from baseline to Day 10 in multi-dose groups.
  Number of Participants with Treatment-Related Adverse Events following administration of UP-818-CC injection.

SECONDARY OUTCOMES:
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (maximum observed drug concentration) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to test the concentration of UP-818-CC and get maximum observed drug concentration.
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (area under the curve) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get area under the curve .
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (time to reach maximum drug concentration) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get time to reach maximum drug concentration.
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (area under the drug-time curve at 0 to infinity time) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get area under the drug-time curve at 0 to infinity time.
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (elimination half-life) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get elimination half-life.
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (clearance rate) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get the clearance rate.
Plasma pharmacokinetic (PK) parameters of UP-818-CC injection (apparent volume of distribution) | Up to 72 hours
  Blood samples will be collected before and up to 72 hours after the administration to get apparent volume of distribution.
Urine pharmacokinetic parameters of UP-818-CC following a single-dose and multiple-doses of UP-818-CC injection (the drug concentration). | Up to 72 hours
  For PK analysis, urine samples will be collected before and up to 72 hours after the administration of UP-818-CC to determine UP-818-CC urine concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The result of this trial has no plan to be published in International Committee of Medical Journal.